CLINICAL TRIAL: NCT04907695
Title: A Prospective Comparison of the Disposable I-view Versus the Durable Video Laryngoscopes in the Emergency Department
Brief Title: Comparing iView Video Laryngoscope in the Emergency Department
Status: Completed | Type: Observational
Sponsor: Brooke Army Medical Center (U.S. Federal Agency)
Collaborators: University of Colorado, Denver (Other)
Responsible Party: Principal Investigator, Steven Schauer, Physician Scientist, Brooke Army Medical Center
Other Study IDs: H-21-022
Record Dates: First submitted 2021-05-10; First posted 2021-06-01 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Intubation; Difficult or Failed; Airway Obstruction
Keywords: Video laryngoscopy; Reusable Video Laryngoscopy devices
MeSH Terms: conditions — Airway Obstruction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Video Laryngoscopy: Seeking all patients undergoing intubation for which the clinician chooses to use Video Laryngoscopy. The participants will undergo intubation with the investigators chosen device.
  Interventions: Device: I View Video Laryngoscope https://www.intersurgical.com/content/files/108253/-1977057700

INTERVENTIONS:
Device: I View Video Laryngoscope https://www.intersurgical.com/content/files/108253/-1977057700 — All intubations will be performed at the direction of the attending clinician. The decision to intubate is based purely on clinical factors by the primary team. The decision to use VL device will be at the direction of the clinical team. No patient will be recruited specific for this procedure.
  Other Names: GlideScope 00879123006400; Storz C-Mac 04048551409381

SUMMARY:
The US Military is rapidly transitioning into preparing for multi-domain operations. Previous data demonstrates that the most common airway replaced in the prehospital combat setting is endotracheal intubation. Previous studies have suggested that video laryngoscopy (VL) is superior to direct laryngoscopy (DL), which is most prominently noted in the office users . However, the current durable equipment video laryngoscopes are very expensive and cost prohibitive for dispersion around the battlefield. The i-view is a novel video laryngoscope that is marketed for VL and is inexpensive and disposable. Both the durable VL and the i-view are already in use in our emergency department (ED). The investigators are also already collecting data using these devices as part of an approved protocol for an airway registry. The investigators are seeking to utilizing a clinical rotating protocol to compare these two devices in the emergency department.

DETAILED DESCRIPTION:
OBJECTIVE:

The investigators are seeking to implement a clinical rotating protocol in which the investigators will use alternating months for which VL device is to be used comparing the i-view to the reusable devices within our department.

The investigators are seeking to answer the following questions:

1. Does the i-view have similar first pass success rates compared to the reusable VL devices (e.g. GlideScope, C-Mac)?
2. Does the i-view have similar attempts required for placement compared to the reusable VL devices?

SUBJECT POPULATION:

The investigators are seeking all patients undergoing intubation for which the clinician chooses to use VL.

NUMBER OF STUDY RECORDS:

The investigators are seeking all encounters for which a VL intubation happens over the course of one years. Our limit will be based on the number of times the procedure occurs.

INCLUSION CRITERIA:

The investigators are seeking any encounter for which the patient undergoes VL intubation as part of routine clinical care.

SAMPLE SIZE ESTIMATION:

A power analysis in SAS version 9.4 (SAS Institute, Cary, NC) indicated that a total sample of 122 would be needed to find that the i-view is non-inferior to the reusable VL if the expected outcome rate (proportion of patients experiencing first-pass success) for the i-view is 87%, the expected outcome rate for the reusable VL is 92%, the noninferiority margin is 5%, power is 80%, and alpha is 5%.

DATA ANALYSIS:

The investigators will use the farrington-Manning score test for non-inferiority to test the first two hypotheses (that the i-view has a non-inferior proportion of patients experiencing hypoxic events, and that the i-view has a non-inferior first-pass success rate compared to the reusable VL devices). The farrington-Manning score test computes the proportion (risk) difference and 90% confidence interval (for a one-sided test) with regards to a predetermined non-inferiority limit. The investigators will use pairwise deletion to handle missing data points (i.e., will only exclude observations if missing data relevant to the specific analysis). Moreover, the investigators may perform regression modeling to adjust for confounders. The investigators performed all statistical analysis using Microsoft Excel (version 10, Redmond, Washington) and JMP Statistical Discovery from SAS (version 13, Cary, NC) or another available commercial software package. The investigators will present continuous variables as means and 95% confidence intervals, non-parametric continuous variables and ordinal variables as medians and interquartile ranges, and nominal variables as percentages and numbers. Significance will be set at p=0.05. The investigators will compare binomial variables using the Chi-square test, normally distributed continuous variables using the Student's t-test, and non-parametric and ordinal variables using the Wilcoxon Rank sum test.

ELIGIBILITY:
Inclusion Criteria:

* We are seeking any encounter for which the patient undergoes VL intubation as part of routine clinical care.

Exclusion Criteria:

* No intubation will be excluded so long as VL is used.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: We are seeking all patients undergoing intubation for which the clinician chooses to use VL.
Sampling Method: Non-Probability Sample
Enrollment: 168 (Actual)
Dates: Start 2021-06-23 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Intubation first-pass success rate | Peri-procedural
  First-pass success between the i-view and the durable VL devices.

CONTACTS AND LOCATIONS:
Overall Officials: Steven G Schauer, DO, Principal Investigator — U.S. Army Institute of Surgical Research
Locations (2):
- United States (2):
  - University of Colorado-Denver, Denver, Colorado
  - Brooke Army Medical Center, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] April MD, Arana A, Pallin DJ, Schauer SG, Fantegrossi A, Fernandez J, Maddry JK, Summers SM, Antonacci MA, Brown CA 3rd; NEAR Investigators. Emergency Department Intubation Success With Succinylcholine Versus Rocuronium: A National Emergency Airway Registry Study. Ann Emerg Med. 2018 Dec;72(6):645-653. doi: 10.1016/j.annemergmed.2018.03.042. Epub 2018 May 7. PMID 29747958
- [Result] April MD, Schauer SG, Brown Rd CA, Ng PC, Fernandez J, Fantegrossi AE, Maddry JK, Summers S, Sessions DJ, Barnwell RM, Antonacci M. A 12-month descriptive analysis of emergency intubations at Brooke Army Medical Center: a National Emergency Airway Registry study. US Army Med Dep J. 2017 Oct-Dec;(3-17):98-104. PMID 29214627
- [Result] Eastridge BJ, Hardin M, Cantrell J, Oetjen-Gerdes L, Zubko T, Mallak C, Wade CE, Simmons J, Mace J, Mabry R, Bolenbaucher R, Blackbourne LH. Died of wounds on the battlefield: causation and implications for improving combat casualty care. J Trauma. 2011 Jul;71(1 Suppl):S4-8. doi: 10.1097/TA.0b013e318221147b. PMID 21795876
- [Result] Eastridge BJ, Mabry RL, Seguin P, Cantrell J, Tops T, Uribe P, Mallett O, Zubko T, Oetjen-Gerdes L, Rasmussen TE, Butler FK, Kotwal RS, Holcomb JB, Wade C, Champion H, Lawnick M, Moores L, Blackbourne LH. Death on the battlefield (2001-2011): implications for the future of combat casualty care. J Trauma Acute Care Surg. 2012 Dec;73(6 Suppl 5):S431-7. doi: 10.1097/TA.0b013e3182755dcc. PMID 23192066
- [Result] Deakin CD, King P, Thompson F. Prehospital advanced airway management by ambulance technicians and paramedics: is clinical practice sufficient to maintain skills? Emerg Med J. 2009 Dec;26(12):888-91. doi: 10.1136/emj.2008.064642. PMID 19934141
- [Result] Liao CC, Liu FC, Li AH, Yu HP. Video laryngoscopy-assisted tracheal intubation in airway management. Expert Rev Med Devices. 2018 Apr;15(4):265-275. doi: 10.1080/17434440.2018.1448267. Epub 2018 Mar 12. PMID 29505333
- [Result] Pott LM, Murray WB. Review of video laryngoscopy and rigid fiberoptic laryngoscopy. Curr Opin Anaesthesiol. 2008 Dec;21(6):750-8. doi: 10.1097/ACO.0b013e3283184227. PMID 18997526
- [Result] Rai MR, Dering A, Verghese C. The Glidescope system: a clinical assessment of performance. Anaesthesia. 2005 Jan;60(1):60-4. doi: 10.1111/j.1365-2044.2004.04013.x. PMID 15601274
- [Result] Serocki G, Bein B, Scholz J, Dorges V. Management of the predicted difficult airway: a comparison of conventional blade laryngoscopy with video-assisted blade laryngoscopy and the GlideScope. Eur J Anaesthesiol. 2010 Jan;27(1):24-30. doi: 10.1097/EJA.0b013e32832d328d. PMID 19809328
- [Result] Schauer SG, Davis WT, Johnson MD, Escandon MA, Uhaa N, Maddry JK, Naylor JF, Van Arnem KA, April MD. A Prospective Assessment of a Novel, Disposable Video Laryngoscope With Physician Assistant Trainees Using a Synthetic Cadaver Model. Mil Med. 2022 May 3;187(5-6):e572-e576. doi: 10.1093/milmed/usaa537. PMID 33289834
- [Result] April MD, Arana A, Reynolds JC, Carlson JN, Davis WT, Schauer SG, Oliver JJ, Summers SM, Long B, Walls RM, Brown CA 3rd; NEAR Investigators. Peri-intubation cardiac arrest in the Emergency Department: A National Emergency Airway Registry (NEAR) study. Resuscitation. 2021 May;162:403-411. doi: 10.1016/j.resuscitation.2021.02.039. Epub 2021 Mar 5. PMID 33684505
- See also: GlideScope — http://accessgudid.nlm.nih.gov/devices/00879123006400
- See also: Storz C-Mac — http://accessgudid.nlm.nih.gov/devices/04048551409381

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-08): https://cdn.clinicaltrials.gov/large-docs/95/NCT04907695/Prot_SAP_000.pdf